CLINICAL TRIAL: NCT04085588
Title: Low Dose Ketamine Infusion for Postoperative Analgesia After Total Knee Arthroplasty: Optimum Dose to Reduce Morphine Consumption
Brief Title: Low Dose Ketamine Infusion for Postoperative Analgesia After Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Selim Turhanoglu, Professor Doctor, Mustafa Kemal University
Other Study IDs: 15.04.2019-07
Record Dates: First submitted 2019-09-05; First posted 2019-09-11 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain
Keywords: Pain; analgesia; Postoperative; Ketamine; Morphine
MeSH Terms: conditions — Pain, Postoperative; Pain; Agnosia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group 1: All patients were revived spinal anesthesia with 3 mL marcaine 0.5% and after surgery a 2 mg bolus morphine PCA pump was connected to them.
  Before the skin incision, when sensorial block reached T10 dermatome level 2 μg / kg / min ketamine was started in Group 1. By the end of the operation ketamine infusion was reduced to 1 μg / kg / min.
- Group 2: All patients were revived spinal anesthesia with 3 mL marcaine 0.5% and after surgery a 2 mg bolus morphine PCA pump was connected to them.
  Before the skin incision, when sensorial block reached T10 dermatome level 4 μg / kg / min ketamine was started . By the end of the operation ketamine infusion was reduced to 2 μg / kg /min and continued.
- Group 3: All patients were revived spinal anesthesia with 3 mL marcaine 0.5% and after surgery a 2 mg bolus morphine PCA pump was connected to them.
  Before the skin incision, when sensorial block reached T10 dermatome level 6 μg / kg / min ketamine was started . By the end of the operation ketamine infusion was reduced to 3 μg / kg /min and continued.

SUMMARY:
This study evaluates continous infusion of low-dose ketamine during intraoperative and postoperative periods at three different doses to provide postoperative analgesia in total knee arthroplasty cases. Patients enrolled randomly into one of 2, 4, 6 μg / kg / min perioperative ketamine groups. All groups were given spinal anesthesia and intravenous patient controlled anesthesia. Ketamine was started when sensorial block reached T10 dermatome level before the skin incision. By the end of the operation, in all groups, ketamine infusions were reduced by half doses. Intravenous patient-controlled analgesia device was set to 2 mg bolus morphine with no basal infusion for 48 hours during the postoperative period.

DETAILED DESCRIPTION:
Multimodal analgesia, which involves the administration of two or more analgesic agents targeting different levels of pain pathways, is used to improve pain control while also to reduce opioid use and related side effects. Pain can be treated at various neurophysiological levels, including peripheral, spinal and cortical targets. One of the agents used in the multimodal analgesia technique is ketamine.

Ketamine acts on the central nervous system (CNS) and has local anesthetic effect. Ketamine is an N-methyl D-Aspartate (NMDA) receptor antagonist, which appears to be the main mechanism of anesthetic and analgesic action at CNS and spinal cord receptors. Other mechanisms of action of ketamine include the interaction with opioid receptors, particularly mu and kappa receptors. Another effect is that it has local anesthetic effect in high doses. Studies have shown that ketamine is an effective agent in the treatment of postoperative pain. Continuous infusion of low-dose ketamine after total knee arthroplasty significantly reduced morphine consumption, and provided early rehabilitation without increasing side effects. However, when these studies are considered, there is no information about the optimal dose of ketamine that reduces opioid consumption at the highest level.

In our study, continuous infusion of low-dose ketamine at different doses was planned to provide postoperative analgesia. Therefore, our first aim in this study was to find out the optimal dose that reduced morphine consumption for postoperative analgesia after TKA with continuous ketamine infusion at different doses. The secondary objectives are to evaluate early and late period pain, side effects, length of hospital stay, patient satisfaction, and recovery.

ELIGIBILITY:
Inclusion Criteria:

• ASA I-Ⅲ female patients scheduled for unilateral total knee arthroplasty

Exclusion Criteria:

* Patients younger than 18 years of age
* ASA Ⅳ and above patients
* Having previous knee surgery on the same side
* Patients with allergies to drugs to be used in the study
* Contraindication for spinal anesthesia
* Body mass index 40 kg / m2 and above patients
* Opioid tolerance
* Patients with neurological or psychiatric disorders
* Patients who do not have the ability to use patient controlled analgesia device

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Being female or male can make difference in pain sensitivity and analgesic response. To facilitate of interpretation the results, only one gender (females) was included in the study.
Study Population: unilateral total knee arthroplasty cases
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Optimal dose of Ketamine to reduce morphine consumption | 48 hours from the operation
  Ketamine infusions 2μg 4μg and 6μg / kg / min will be started preoperatively in group 1, 2 and 3 respectively when sensory block level reaches T10 after spinal anesthesia, and they will be reduced by half by the end of the operation. Ketamine infusion will be continued for 48 hours postoperatively.

SECONDARY OUTCOMES:
Early and late period pain | 3 months from the operation
  The pain status of the patients at rest and in motion with 100 mm visual pain scale (VAS) (0= no pain and 100 = intolerable pain) will be evaluated and recorded preoperative and postoperative at 2nd, 6th, 12th, 24th and 48th hours.and after 3 months
side effects, | 3 months
  Nausea, vomiting, itching, respiratory depression, hallucination and diplopia
length of hospital stay | 3 months
  Hospital stay (as day) required for active knee flexion to 90 degrees (measured with goniometer) will be recorded.
patient satisfaction | 3 months
  5 point likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Selim Turhanoglu, M.D., Study Director — Mustafa Kemal University, Medical School, 31100 Hatay, Turkey
Locations (1):
- Mustafa Kemal University Medical School, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Sharing data have not been discussed among the investigators yet.

REFERENCES:
- [Result] Memtsoudis SG, Poeran J, Zubizarreta N, Cozowicz C, Morwald EE, Mariano ER, Mazumdar M. Association of Multimodal Pain Management Strategies with Perioperative Outcomes and Resource Utilization: A Population-based Study. Anesthesiology. 2018 May;128(5):891-902. doi: 10.1097/ALN.0000000000002132. PMID 29498951
- [Result] Schmid RL, Sandler AN, Katz J. Use and efficacy of low-dose ketamine in the management of acute postoperative pain: a review of current techniques and outcomes. Pain. 1999 Aug;82(2):111-125. doi: 10.1016/S0304-3959(99)00044-5. PMID 10467917
- [Result] Adam F, Chauvin M, Du Manoir B, Langlois M, Sessler DI, Fletcher D. Small-dose ketamine infusion improves postoperative analgesia and rehabilitation after total knee arthroplasty. Anesth Analg. 2005 Feb;100(2):475-480. doi: 10.1213/01.ANE.0000142117.82241.DC. PMID 15673878
- [Result] Aveline C, Gautier JF, Vautier P, Cognet F, Hetet HL, Attali JY, Leconte V, Leborgne P, Bonnet F. Postoperative analgesia and early rehabilitation after total knee replacement: a comparison of continuous low-dose intravenous ketamine versus nefopam. Eur J Pain. 2009 Jul;13(6):613-9. doi: 10.1016/j.ejpain.2008.08.003. Epub 2008 Sep 14. PMID 18793861
- [Result] Pai A, Heining M. Ketamine. Continuing Education in Anaesthesia, Critical Care and Pain 2007; Volume 7,Number 2.